CLINICAL TRIAL: NCT03552874
Title: The Comparison of Pulmonary and Upper Extremity Functions Between Children With Duchenne Muscular Dystrophy and Healthy Peers
Brief Title: Pulmonary and Upper Limb Functions in Duchenne Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Numan Bulut, Department of Physiotherapy and Rehabilitation, Principal Investigator, Research Assistant, Hacettepe University
Other Study IDs: GO 16/773
Record Dates: First submitted 2018-05-25; First posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Duchenne Muscular Dystrophy; Upper Limb Function; Respiratory Function Test
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient Group: Children whose ages between 5-10 years with Duchenne Muscular Dystrophy.
  Interventions: Other: The Performance of Upper Limb Questionnaire (PUL)
- Healthy Group: Healthy peers
  Interventions: Other: The Performance of Upper Limb Questionnaire (PUL)

INTERVENTIONS:
Other: The Performance of Upper Limb Questionnaire (PUL)
  Other Names: Pulmonary Function Test (PFT)

SUMMARY:
Although it is known that the functions of pulmonary and upper limb is affected in late stage of Duchenne Muscular Dystrophy (DMD) negatively, the investigators do not have clear information about its early stage. The aim of this study was to investigate the differences in pulmonary and upper limb functions between children with DMD in early stage and healthy peers.

ELIGIBILITY:
Inclusion Criteria:

children with DMD was;

* age between 5-10 years
* being on treatment with corticosteroids for more than 6 months
* being at Level I according to Brooke Upper and Lower Extremity Classification Systems

Healthy peers;

* age between 5-10 years
* not having any diagnosed disease

Exclusion Criteria:

• Children has undergo surgery and disease affect upper extremity or pulmonary function in last six months.

Ages: 5 Years to 10 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — This study is gender based because Duchenne Muscular Dystrophy is only seen in males.
Study Population: Fourty seven participants including 31 children with DMD and 16 healthy peers were included
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function Test (PFT) | 5 minutes
  The pulmonary function tests of the participants were evaluated with a spirometry. The child was asked to perform the spirometric tests for three times with maximum effort. The child was motivated before each attempt for stronger and longer expiration.The result of Pulmonary function Test were recorded.
The Performance Upper Limb (PUL) | 15 minutes
  Upper limb functions of participants were evaluated with The Performance of Upper Limb (PUL) scale. This scale, which was shown to be reliable in DMD, has 22 items in total. It consists of 3 different levels of function: high, mid, and distal. PUL also has four items determining timed performance.

IPD SHARING:
Plan to Share IPD: No